CLINICAL TRIAL: NCT00000459
Title: Dietary Intervention Study in Children (DISC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 48; U01HL037947 (NIH); U01HL037948 (NIH); U01HL037954 (NIH); U01HL037962 (NIH); U01HL037966 (NIH); U01HL037975 (NIH); U01HL038110 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2005-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypercholesterolemia
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypercholesterolemia | interventions — Diet, Fat-Restricted

INTERVENTIONS:
Behavioral: diet, fat-restricted

SUMMARY:
To assess the feasibility, acceptability, efficacy, and safety of dietary intervention in free-living children ages 8-10 with elevated low density lipoprotein cholesterol levels.

DETAILED DESCRIPTION:
BACKGROUND:

Several lines of evidence provided the rationale for intervening in children. A large body of autopsy and pathologic evidence had accumulated showing that atherosclerosis, including fatty streaks, increased surface involvement, and advanced microscopic lesions, began in childhood. Blood cholesterol levels tracked from childhood to adulthood, with tracking correlations ranging from .6 to .8. Therefore, a high proportion of children with high levels of cholesterol have high levels as adults. Family clustering of risk factors had also been reported. Studies showed 2-3 times increased prevalence of coronary heart disease in adult relatives of children with high cholesterol compared to children with normal cholesterol, and 2.2 times increased prevalence in high cholesterol in children who had a parent or grandparent with premature coronary heart disease compared with children who did not have a family history of premature heart disease. Finally, there was high likelihood that environmental influences on coronary heart disease risk factors had their behavioral antecents in childhood. Thus, dietary habits which contributed toward elevated blood cholesterol levels were likely to have developed early in life, and it was hoped that behavioral change achieved during childhood was likely to persist into adulthood.

Although numerous studies had shown that dietary modification could lower blood cholesterol levels in adults, only a few studies had shown this effect in children, and none were long-term. Furthermore, the impact on long-term growth and development in children had not been studied. Concerns were raised about the safety of cholesterol-lowering diets in children, particularly during peak growing years. These concerns included possible deficits in growth and nutrient adequacy, and potential adverse psychological effects. This paucity of data was a potential barrier to active prevention measures. To fill this gap in knowledge, the DISC trial, a randomized, controlled clinical trial, tested the efficacy and safety of long-term dietary intervention for reduction of serum LDL-C levels in children during puberty.

DESIGN NARRATIVE:

In the feasibility study, children of both sexes, ages 8 to 10 at baseline starting in 1987, were randomized to either a control group or to a usual care group for whom more intensive dietary intervention for the child and the family was directed. The feasibility study lasted 16 months. The full-scale trial began in December 1988 with the randomization of a total of 663 children. At baseline, mean LDL-C levels, nutrient intakes, anthropometric measurements, nutritional biochemical levels, and psychosocial measures were similar in the two groups. The intervention group was assigned to a series of group and individual sessions to teach the children and their families to follow a diet containing 28 percent of calories as total fat, dietary cholesterol intake less than 75 mg/1000 kcal, and up to 9% of calories from polyunsaturated fat. The diets were designed to meet nutritional requirements of growing children. The usual care group was provided a packet of general dietary information only. The primary efficacy outcome was a difference in changes in LDL-C levels between the two groups at 36 months. Primary safety endpoints were change in height and serum ferritin levels. Secondary safety outcomes included serum zinc, retinol, albumin levels, red blood cell folate, ratio of LDL-C to high-density lipoprotein cholesterol, sexual maturation, cognitive development, and psychosocial assessments. Recruitment was completed in July 1990. Intervention and follow-up was extended until 1997 when the participants were on average 17 years old. Data analysis continued through January 1999.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Children, ages 8 to 10, with elevated LDL-C levels.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1986-12; Study Completion 1999-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Barton — Maryland Medical Research Institute

REFERENCES:
- [Background] Van Horn LV, Gernhofer N, Moag-Stahlberg A, Farris R, Hartmuller G, Lasser VI, Stumbo P, Craddick S, Ballew C. Dietary assessment in children using electronic methods: telephones and tape recorders. J Am Diet Assoc. 1990 Mar;90(3):412-6. PMID 2307817
- [Background] Dietary intervention study in children (DISC) with elevated low-density-lipoprotein cholesterol. Design and baseline characteristics. DISC Collaborative Research Group. Ann Epidemiol. 1993 Jul;3(4):393-402. doi: 10.1016/1047-2797(93)90067-e. PMID 8275216
- [Background] van Horn LV, Stumbo P, Moag-Stahlberg A, Obarzanek E, Hartmuller VW, Farris RP, Kimm SY, Frederick M, Snetselaar L, Liu K. The Dietary Intervention Study in Children (DISC): dietary assessment methods for 8- to 10-year-olds. J Am Diet Assoc. 1993 Dec;93(12):1396-403. doi: 10.1016/0002-8223(93)92241-o. PMID 8245373
- [Background] Hartmuller VW, Snetselaar L, Van Horn L, et al: Creative Approaches to Cholesterol-Lowering Used in the Dietary Intervention Study in Children (DISC). Top Clin Nutr, 10:71-78, 1994.
- [Background] Efficacy and safety of lowering dietary intake of fat and cholesterol in children with elevated low-density lipoprotein cholesterol. The Dietary Intervention Study in Children (DISC). The Writing Group for the DISC Collaborative Research Group. JAMA. 1995 May 10;273(18):1429-35. doi: 10.1001/jama.1995.03520420045036. PMID 7723156
- [Background] Stevens VJ, Obarzanek E, Franklin FA, et al for the DISC Collaborative Research Group. Dietary Intervention Study in Children (DISC): intervention design and participation. J Nutr Educ 1995;27:133-140.
- [Background] Luepker RV. Reducing blood cholesterol levels in children. What have we learned from the DISC study? JAMA. 1995 May 10;273(18):1461-2. No abstract available. PMID 7723162
- [Background] Simons-Morton DG, Hunsberger SA, Van Horn L, Barton BA, Robson AM, McMahon RP, Muhonen LE, Kwiterovich PO, Lasser NL, Kimm SY, Greenlick MR. Nutrient intake and blood pressure in the Dietary Intervention Study in Children. Hypertension. 1997 Apr;29(4):930-6. doi: 10.1161/01.hyp.29.4.930. PMID 9095079
- [Background] Obarzanek E, Hunsberger SA, Van Horn L, Hartmuller VV, Barton BA, Stevens VJ, Kwiterovich PO, Franklin FA, Kimm SY, Lasser NL, Simons-Morton DG, Lauer RM. Safety of a fat-reduced diet: the Dietary Intervention Study in Children (DISC). Pediatrics. 1997 Jul;100(1):51-9. doi: 10.1542/peds.100.1.51. PMID 9200359
- [Background] Kwiterovich PO Jr, Barton BA, McMahon RP, Obarzanek E, Hunsberger S, Simons-Morton D, Kimm SY, Friedman LA, Lasser N, Robson A, Lauer R, Stevens V, Van Horn L, Gidding S, Snetselaar L, Hartmuller VW, Greenlick M, Franklin F Jr. Effects of diet and sexual maturation on low-density lipoprotein cholesterol during puberty: the Dietary Intervention Study in Children (DISC). Circulation. 1997 Oct 21;96(8):2526-33. doi: 10.1161/01.cir.96.8.2526. PMID 9355889
- [Background] Reimers TM, Brown KM, Van Horn L, Stevens V, Obarzanek E, Hartmuller VW, Snetselaar L, von Almen TK, Chiostri J. Maternal acceptability of a dietary intervention designed to lower children's intake of saturated fat and cholesterol: the Dietary Intervention Study in Children (DISC). J Am Diet Assoc. 1998 Jan;98(1):31-4. doi: 10.1016/s0002-8223(98)00010-8. PMID 9434647
- [Background] Berg-Smith SM, Stevens VJ, Brown KM, Van Horn L, Gernhofer N, Peters E, Greenberg R, Snetselaar L, Ahrens L, Smith K. A brief motivational intervention to improve dietary adherence in adolescents. The Dietary Intervention Study in Children (DISC) Research Group. Health Educ Res. 1999 Jun;14(3):399-410. doi: 10.1093/her/14.3.399. PMID 10539230
- [Background] Obarzanek E, Kimm SY, Barton BA, Van Horn L L, Kwiterovich PO Jr, Simons-Morton DG, Hunsberger SA, Lasser NL, Robson AM, Franklin FA Jr, Lauer RM, Stevens VJ, Friedman LA, Dorgan JF, Greenlick MR; DISC Collaborative Research Group. Long-term safety and efficacy of a cholesterol-lowering diet in children with elevated low-density lipoprotein cholesterol: seven-year results of the Dietary Intervention Study in Children (DISC). Pediatrics. 2001 Feb;107(2):256-64. doi: 10.1542/peds.107.2.256. PMID 11158455
- [Background] Lauer RM, Obarzanek E, Hunsberger SA, Van Horn L, Hartmuller VW, Barton BA, Stevens VJ, Kwiterovich PO Jr, Franklin FA Jr, Kimm SY, Lasser NL, Simons-Morton DG. Efficacy and safety of lowering dietary intake of total fat, saturated fat, and cholesterol in children with elevated LDL cholesterol: the Dietary Intervention Study in Children. Am J Clin Nutr. 2000 Nov;72(5 Suppl):1332S-1342S. doi: 10.1093/ajcn/72.5.1332s. PMID 11063475
- [Background] Lavigne JV, Brown KM, Gidding S, Evans M, Stevens VJ, von Almen TK, Ewart C, Weil C. A cholesterol-lowering diet does not produce adverse psychological effects in children: three-year results from the dietary intervention study in children. Health Psychol. 1999 Nov;18(6):604-13. doi: 10.1037//0278-6133.18.6.604. PMID 10619534
- [Derived] Jung S, Goloubeva O, Hylton N, Klifa C, LeBlanc E, Shepherd J, Snetselaar L, Van Horn L, Dorgan JF. Intake of dietary carbohydrates in early adulthood and adolescence and breast density among young women. Cancer Causes Control. 2018 Jul;29(7):631-642. doi: 10.1007/s10552-018-1040-1. Epub 2018 May 25. PMID 29802491
- [Derived] Bertrand KA, Baer HJ, Orav EJ, Klifa C, Kumar A, Hylton NM, LeBlanc ES, Snetselaar LG, Van Horn L, Dorgan JF. Early Life Body Fatness, Serum Anti-Mullerian Hormone, and Breast Density in Young Adult Women. Cancer Epidemiol Biomarkers Prev. 2016 Jul;25(7):1151-7. doi: 10.1158/1055-9965.EPI-16-0185. Epub 2016 May 9. PMID 27197299
- [Derived] Jung S, Egleston BL, Chandler DW, Van Horn L, Hylton NM, Klifa CC, Lasser NL, LeBlanc ES, Paris K, Shepherd JA, Snetselaar LG, Stanczyk FZ, Stevens VJ, Dorgan JF. Adolescent endogenous sex hormones and breast density in early adulthood. Breast Cancer Res. 2015 Jun 4;17(1):77. doi: 10.1186/s13058-015-0581-4. PMID 26041651
- [Derived] Uchino R, Isayama H, Tsujino T, Sasahira N, Ito Y, Matsubara S, Takahara N, Arizumi T, Toda N, Mohri D, Togawa O, Yagioka H, Yanagihara Y, Nakajima K, Akiyama D, Hamada T, Miyabayashi K, Mizuno S, Kawakubo K, Kogure H, Sasaki T, Yamamoto N, Nakai Y, Hirano K, Tada M, Koike K. Results of the Tokyo trial of prevention of post-ERCP pancreatitis with risperidone-2: a multicenter, randomized, placebo-controlled, double-blind clinical trial. Gastrointest Endosc. 2013 Dec;78(6):842-850. doi: 10.1016/j.gie.2013.06.028. Epub 2013 Jul 30. PMID 23910063
- [Derived] Dorgan JF, Liu L, Barton BA, Deshmukh S, Snetselaar LG, Van Horn L, Stevens VJ, Robson AM, Lasser NL, Himes JH, Shepherd JA, Pourfarzib R, Pettee Gabriel K, Kriska A, Kwiterovich PO Jr. Adolescent diet and metabolic syndrome in young women: results of the Dietary Intervention Study in Children (DISC) follow-up study. J Clin Endocrinol Metab. 2011 Dec;96(12):E1999-2008. doi: 10.1210/jc.2010-2726. Epub 2011 Oct 12. PMID 21994964
- [Derived] Kerver JM, Gardiner JC, Dorgan JF, Rosen CJ, Velie EM. Dietary predictors of the insulin-like growth factor system in adolescent females: results from the Dietary Intervention Study in Children (DISC). Am J Clin Nutr. 2010 Mar;91(3):643-50. doi: 10.3945/ajcn.2009.28205. Epub 2010 Jan 20. PMID 20089725